CLINICAL TRIAL: NCT05788874
Title: Comparative Study of 18F-FAPI and 18F-FDG PET/CT for Gastrointestinal Cancer
Brief Title: Study of 18F-FAPI Applied to Gastrointestinal Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF-CRF-2022-021
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 18F-FDG
  Interventions: Diagnostic Test: 18F-FAPI and 18F-FDG PET/CT
- 18F-FAPI
  Interventions: Diagnostic Test: 18F-FAPI and 18F-FDG PET/CT

INTERVENTIONS:
Diagnostic Test: 18F-FAPI and 18F-FDG PET/CT — 18F-FAPI and 18F-FDG PET/CT for gastrointestinal cancer

SUMMARY:
Comparison of tumor volume, number, and SUVmax of different primary foci (gastric, duodenal, and colon cancer), lymph node metastases (neck and supraclavicular, mediastinal, abdominal, and pelvic), and distant metastases (brain, lung, liver, bone, pleura, and peritoneum) detected by 18F-FAPI versus 18F-FDG PET/CT imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients with high clinical suspicion of gastrointestinal tumor and negative 18F-FDG at first diagnosis
* Post-treatment patients with high clinical suspicion of recurrence or metastasis and negative 18F-FDG

Exclusion Criteria:

* The diagnosis can be clarified by 18F-FDG PET/CT examination
* The presence of recurrence or metastasis can be clarified by 18F-FDG PET/CT examination

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Patients with high clinical suspicion of gastrointestinal tumor and negative 18F-FDG at first diagnosis
  * Post-treatment patients with high clinical suspicion of recurrence or metastasis and negative 18F-FDG
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
SUVmax | 1 day (During the inspection)
  Measurement of the maximum standardized uptake value of the lesion

IPD SHARING:
Plan to Share IPD: No